CLINICAL TRIAL: NCT06062381
Title: The Effect of Abdominal Massage on the Gastric Residual Volume in Adult Patients Admitted in Intensive Care Unit: A Randomized Controlled Trial
Brief Title: the Effect of Abdominal Massage on the Gastric Residual Volume.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Mahwish Javeed, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GRV RCT 001
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Gastric Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): experimental group will receive abdominal massage of 20 minutes duration for 3 days.
  Interventions: Procedure: Abdominal Massage
- Control Group (No Intervention): control group will receive only routine care

INTERVENTIONS:
Procedure: Abdominal Massage — The intervention period will be 3 days for intervention group. These patients will receive 20 minutes of abdominal massage twice a day, and the interval between two massages will be 2 hours. The outcome variable variable gastric residual volume will be measured every day, before the intervention and 1 hour after the second massage. the GRV will be measured in ml (via feeding syringe) and marked on checklist.
  The abdominal massage technique will consist of five steps based on tensegrity principle.
  The lubricant gel will be used to facilitate the massaging. The patient's position will be supine while going through abdominal massage. The angle between the bed and the patient's head will be 30 to 45 degrees, and the patient's legs will be placed on a pillow. This condition will help to relax the abdominal muscles.
  Arms: Intervention Group

SUMMARY:
The goals of this randomized controlled trial are:

1. To determine the mean gastric residual volume in ICU admitted adult patients before and after intervention.
2. To compare the gastric residual volume between the intervention and control group.

Participants will be randomized in two groups (intervention and control group)

Intervention group:

The intervention period will be 3 days for intervention group. These patients will receive 20 minutes of abdominal massage twice a day, and the interval between two massages will be 2 hours. The outcome variable variable gastric residual volume will be measured every day, before the intervention and 1 hour after the second massage. the GRV will be measured in ml (via feeding syringe) and marked on checklist.

Control group The control group will receive standard/usual care The abdominal massage technique will consist of five steps based on tensegrity principle

DETAILED DESCRIPTION:
Food intolerance is one of the major problems of intensive care unit (ICU) admitted patients, receiving enteral nutrition. An important nursing priority for these patients is the prevention and management of food intolerance. This necessitates the use of techniques and procedures for increasing the rate of gastric emptying, and so enhancing tolerance to this nutritional support modality. Abdominal massage is a method that has shown to improve many digestive functions such as constipation and gastric residual volume (GRV), but a small number of studies have been conducted on NG fed patients in intensive care units, and occasionally, contradictory findings have been found. Furthermore, more studies were recommended to reach a definite conclusion on this intervention. The aim of this study is to determine the effect of abdominal massage on the gastric residual volume in patients hospitalized in intensive care units in a tertiary care hospital, Lahore. It is hypothesized that ICU admitted patients who will receive abdominal massage will have a difference in gastric residual volume than patients who will not.

Study Design A randomized controlled trial (RCT). Study setting The study will be conducted at Intensive care units of Jinnah Hospital, Lahore. Study Population Patients having nasogastric tube (NGT) for feeding and admitted in ICU with GCS below 7.

Sample size A sample size of 34 patients is calculated by using the formula of comparing means between two group and by taking power of study 80%, confidence level 95% ,mean gastric residual volume of intervention group 97.30 ml, mean gastric residual volume of control group 143.46 ml, standard deviation of gastric residual volume of intervention group 54.06 ml and standard deviation of gastric residual volume of control group = 39.93 ml.

Sampling technique patients will first be selected by non-probability convenient sampling. Then patients will be randomized into two groups by lottery method (17 patients in each group).

Data will be collected by using a researcher-designed checklist which will consist of two parts:

Demographic characteristics and medical data Gastric residual volume (GRV) monitoring The intervention period will be 3 days for intervention group. These patients will receive 20 minutes of abdominal massage twice a day, and the interval between two massages will be 2 hours. Every day, before the intervention and 1 hour after the second massage, the GRV will be measured I ml (via feeding syringe) and marked on checklist. The abdominal massage technique will consist of five steps based on tensegrity principle.

Data will be analyzed by using statistical package for social sciences (SPSS) version 24. Descriptive statistics (frequency, percentage, mean and standard deviation) will be used to describe the characteristics of study population. Chi square test will be used to examine the demographic information of the two groups based on qualitative variables. Independent t test will be used to compare the mean of the total GRV in both groups before and after intervention. The significance level of the tests will be considered at <0.05 Findings of this study will provide base line data about the effectiveness of abdominal massage among adult critically ill patients' gastric residual volume. This procedure can be considered as a care method to improve nutrition status in patients hospitalized in these units. This inexpensive and complementary nursing therapy will be suggested to add in standard ICU nursing care practices for decreasing gastric residual volume and fulfilling required calorie intake, decreasing risk of complications and hospital stay and improving healing.

ELIGIBILITY:
Inclusion Criteria:

* patients having NG tube (for check the GRV).
* glasgow coma scale less than 7 (because usually these patients need gavage)
* patients having age 18-60 years.

Exclusion Criteria:

* Patients receiving pro-kinetic medications (to avoid interfering with the massage effects)
* Patients having abdominal radiotherapy during last 6 weeks.
* Patients with abdominal aortic aneurysm and undergoing radiotherapy
* Patients having abdominal surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Gastric Residual Volume | before and after intervention ( 3 hours duration)
  Gastric residual volume will be measured in ml by aspiration of gastric contents.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No